CLINICAL TRIAL: NCT02131116
Title: An Integrated Metacognitive Approach to Improve Insight and Outcomes in Early Psychosis
Brief Title: Integrated Metacognitive Therapy in First Episode Psychosis
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jenifer Vohs, Clinical Psychologist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1401410369
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: schizophrenia; schizophreniform disorder; schizoaffective disorder; cognition; metacognition; insight; first episode psychosis; psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMT (Experimental): Integrated Metacognitive Therapy
  Interventions: Behavioral: Integrated Metacognitive Therapy; Behavioral: Treatment as Usual
- TAU (No Intervention): No intervention group/Treatment as Usual

INTERVENTIONS:
Behavioral: Integrated Metacognitive Therapy — Integrated Metacognitive Therapy
  Arms: IMT
Behavioral: Treatment as Usual — Treatment as Usual
  Other Names: No intervention/Treatment as Usual
  Arms: IMT

SUMMARY:
Insight, or lack of illness awareness, is a prominent and pressing clinical concern in the treatment and recovery of patients with psychotic disorders. Impaired insight results in poor treatment engagement and adherence, more frequent hospitalizations, greater positive and negative symptoms, and poor psychosocial functioning. Addressing these complications early in the disease process may lead to altered illness course with better outcomes. To date, only a small number of nonpharmacological interventions have been developed, none of which adequately address poor insight during the first few years of psychotic illness. Further, presently available therapeutic interventions do not attend to difficulties associated with improved insight, such as depression. The purpose of this investigation is to implement a novel intervention designed to improve insight, metacognition, neurocognition, symptoms, and ultimately overall functioning in persons with early psychosis. The novel intervention will integrate a number of previously established therapeutic approaches, such as metacognitive, narrative, cognitive behavioral and motivational interviewing, and hence be labeled Integrated Metacognitive Therapy (IMT). In order to measure the efficacy of IMT, all subjects will undergo a battery of assessments in each of these domains prior to and following either a novel intervention (N = 10) or treatment as usual (N = 10) for a period of approximately six months. Throughout the study, each IMT session (N = 10, 24 sessions each) will be audio recorded, transcribed, and de-identified to allow for careful ongoing qualitative analyses of potential active and inert ingredients of the approach and ultimately the development of an IMT manual which can then be tested in a larger, more rigorous randomized control trial. This investigation will play an important role in advancing current knowledge about treating insight in early psychosis. Further, it will serve to expand upon the intervention tools available by producing a much needed treatment manual designed specifically to target insight during an illness phase crucial for positive long term outcomes in psychosis.

DETAILED DESCRIPTION:
The National Advisory Mental Health Council recently called for the development of non-pharmacological treatments that identify and target specific disease processes for clinical improvement in schizophrenia and other psychotic illnesses. One such illness process, vital for positive outcomes, is impaired awareness of illness or insight. Insight is often thought of as factual knowledge and acknowledgement of one's illness. More specifically, insight in psychosis has been conceptualized as a multi-dimensional construct, with several independent but overlapping dimensions, such as the ability to appropriately label aberrant mental events (e.g. hallucinations and delusions), recognition of illness, and willingness to engage in treatment. Relative to individuals with other mental illnesses, those with psychotic illness have the most impaired insight, presenting a number of challenges, including: poor treatment engagement and adherence, more frequent hospitalizations, greater positive and negative symptoms, and poor psychosocial functioning. This problem is particularly relevant in early phases of psychotic illness, where there remains a paucity of data. Data that is available has shown decreased insight is associated with increased symptoms and poorer cognitive functioning, both of which have the potential to impact illness course.

Two reasons account for a lack of attention to the development of treatments for insight: i) the lack of an adequate model of the forces which cause and sustain poor insight and ii) a failure to consider an integrated treatment. Without an idea of the processes which sustain poor insight, interventions have been able to offer education about the nature of illness but have not been equipped to respond to the underlying processes that block the emergence of insight in treatment. While earlier literature framed insight as a failure to grasp a specific fact, more recent efforts suggest poor insight is primarily the result of a failure to create a coherent account of the complex events and personal experiences related to a psychiatric illness. These difficulties becoming aware of one's illness may be multi-determined and result from factors including deficits in metacognition, neurocognition, and symptoms.

The development of insight is complex and highly dependent upon metacognitive processes, which have a unique, potentially moderating role. Metacognition involves a range of faculties that allow an individual to form representations of mental states of self and others, which then leads to the formation and revision of thoughts, beliefs, feelings, behaviors, and even individual aspirations. Therapies targeting metacognitive or mentalizing deficits have been successfully implemented for personality disorders, depression and anxiety. In psychotic disorders, decreased metacognitive capacity is thought to result in difficulties identifying the source of one's experiences, such as illness and its consequences. This leads to an inability to perceive the self as an active agent in the world and problems in understanding and acting upon the social cues (emotions and intentions) of others. A recently proposed Integrated Metacognitive therapeutic approach argues that insight will improve as an individual utilizes a constructed narrative to make sense of his or her experiences. In other words, illness and its consequences are understood in an individualized, personally relevant and acceptable way. Importantly, this approach addresses many obstacles to gaining insight not addressed by other approaches, including learning to deal with related emotional pain and depression, loss, and internalized stigma. This view is also consistent with intervention research showing that establishment of personal meaning is important for recovery, and promotes improved function and reduced symptoms. Case studies from our group and others have provided evidence that therapy targeting metacognitive processes is feasible in psychotic disorders and can indeed improve insight and function in persons with chronic schizophrenia. However, this approach has not been tailored to target insight, evaluated or tested in patients in the early phase of psychosis.

In addition to metacognitive deficits, neurocognitive deficits have also been commonly observed in schizophrenia and involve decrements in capacities for attention/vigilance, verbal memory and executive function. Deficits in executive function have been found to predict concurrent and prospective assessments of poorer insight, spurring hypotheses that impairments in executive function leave persons unable to synthesize illness related experiences into a coherent and adequate story about how and why they are ill. Deficits in attention and memory may additionally obscure how historical events are connected to each other. As a whole, neurocognitive deficits may cause difficulties piecing together the individual's experience of illness into a coherent whole resulting in poor insight. Therefore, development of personal narratives using an integrated therapy would allow subjects the opportunity to better understand their illness experience, hence improving insight.

The research presented above suggests that improving insight early in the psychotic disease process would likely result in improved treatment participation, ultimately leading to better outcomes. Motivated by a clear and pressing need to better address illness insight in early psychotic illness and recent positive findings related to doing so, the present investigation serves to test a novel Integrated Metacognitive Therapy (IMT) which targets insight and other important domains in early psychosis. Assuming IMT is successful, ongoing qualitative analysis of IMT sessions will allow for manual development, future randomized control trials, and ultimately treatment dissemination.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age at study entry
* Male or female
* DSM IV-TR Diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder as confirmed by Structured Clinical Interview for DSM-IV-TR (SCID)
* Onset of schizophreniform disorder, schizophrenia, or schizoaffective disorder within the past five years as defined by first medical records documentation of these conditions
* Score of 4 or higher (moderate impairment) on the Positive and Negative Syndrome Scale (PANSS) insight item

Exclusion Criteria:

* History of significant neurological illness or head trauma
* Known IQ < 70 based on medical history
* Current alcohol or drug dependence (excluding nicotine or caffeine) based on the SCID interview.
* Subjects considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 90 days prior to screening

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Insight | 24 weeks
  improved insight as measured by the Scale of Unawareness of Illness
Insight | 24 weeks
  Insight item on the Positive and Negative Syndrome Scale
Insight | 24 weeks
  Beck Cognitive Insight Scale
metacognition | 24 weeks
  Bell Lysaker Emotion Recognition Test
metacognition | 24 weeks
  scores on the the Eyes Test
metacognition | 24 weeks
  scores on the Hinting Test
metacognition | 24 weeks
  Indiana Psychiatric Illness Interview and Metacognitive Assessment Scale),

SECONDARY OUTCOMES:
overall symptomatology | 24 weeks
  Positive and Negative Syndrome Scale
overall symptomatology | 24 weeks
  Liebowitz Social Anxiety Scale
neurocognition | 24 weeks
  Brief Assessment for Cognition in Schizophrenia total score
neurocognition | 24 weeks
  Trail Making Test, Part B
social functioning | 24 weeks
  Quality of Life Scale
social functioning | 24 weeks
  Social Functioning Scale
social functioning | 24 weeks
  Marlow-Crowne Social Desirability Scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana
  - Psychosocial Rehabilitation and Recovery Center, Indianapolis, Indiana